CLINICAL TRIAL: NCT06674577
Title: A Multicenter, Rollover Study to Evaluate the Long-Term Safety and Efficacy of Atacicept
Brief Title: A Rollover Study to Evaluate the Long-Term Safety and Efficacy of Atacicept
Acronym: ORIGIN EXTEND
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Vera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VT-001-0051
Record Dates: First submitted 2024-10-03; First posted 2024-11-05 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-12

CONDITIONS: IgA Nephropathy (IgAN); Renal and Urinary Disorders; Berger Disease
Keywords: IGA Glomerulonephritis; IGA Nephropathy; Iga Nephropathy 1; Immunoglobulin A Nephropathy Nephritis; IGA Type Nephropathy, IGA; renal and urinary disorders; Berger Disease; Berger's Disease
MeSH Terms: conditions — Glomerulonephritis, IGA; Urologic Diseases | interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atacicept 150mg once weekly subcutaneous (SC) injection (Experimental): Other Names:
  VT-001
  Interventions: Drug: Atacicept 150 mg

INTERVENTIONS:
Drug: Atacicept 150 mg — The atacicept drug product is available as a ready to use injection solution in the following prefilled syringe (PFS) that is composed of: *BD Hypak™ SCF™ Barrel Glass barrel 1ml long with staked needle 27G ½" 5B with Rigid Needle Shield BD260 *BD SCF™ Stopper 1ml long W4023 Flurotec

SUMMARY:
The purpose of this study is to collect long-term safety and tolerability data for atacicept in patients with IgAN that completed Vera trial investigating atacicept in IgAN population.

DETAILED DESCRIPTION:
Eligible participants will receive atacicept 150 mg once weekly (QW) self-administered subcutaneously (SC). Participants will be grouped by whether they are restarting atacicept after cessation in the parent study (Group 1: Atacicept Drug Holiday) or are continuing atacicept with no disruption in treatment (Group 2: Continuous Atacicept Treatment). Long-term safety and tolerability of atacicept is assessed by routine clinical and laboratory tests and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study assessments
* Completed the protocol-defined treatment period on treatment in a parent study of atacicept in patients with IgAN
* For Atacicept Drug Holiday Group only: Systolic blood pressure ≤150 mmHg and diastolic blood pressure ≤90mmHg at screening and Day 1
* A participant who was assigned female at birth is eligible if not pregnant (ie, after a confirmed menstrual period, a negative serum pregnancy test at screening and has a negative urine pregnancy test at Day 1), is not breastfeeding (for at least three months prior to screening), and at least one of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP) OR
  * Is a WOCBP who agrees to use a highly effective contraceptive method (ie, has a failure rate of less than 1% per year) at least 7 days prior to enrollment, through 175 days after the last dose of study drug.

Exclusion Criteria:

* Evidence of rapidly progressive glomerulonephritis (loss of ≥50% of eGFR within 3 months of screening)
* For Atacicept Drug Holiday Group only: History of splenectomy
* Known hypersensitivity to atacicept or any component of the formulated atacicept
* For Atacicept Drug Holiday Group only: Major surgery within 6 weeks prior to screening or planned/expected major surgery during the study period (including the safety follow-up period). Major surgery often involves opening one of the major body cavities (abdomen or chest) and/or use of general anesthesia. Types of surgery that have the highest risk include heart or lung, liver, abdomen, or major operations on the bones and joints (eg, hip replacement)
* Clinically significant history of alcohol or drug abuse in the 1 year prior to Day 1 as per Investigator opinion
* Unwillingness or lack of capacity to follow all study procedures
* For Atacicept Drug Holiday Group only: Treatment with other investigational agents within the last 4 weeks or 5 half-lives, whichever is longer, prior to screening
* Evidence of nephrotic syndrome (serum albumin <30g/L in association with UPCR >3.5 mg/mg) within 6 months of screening
* Currently on chronic dialysis, or expected to initiate dialysis within 12 weeks of screening
* Renal or other organ transplantation prior to, or expected during, the study, with the exception of corneal transplants
* Clinically significant or predefined abnormalities per central laboratory tests at screening, meeting any of the criteria: Clinical evidence of immunosuppression and/or hypogammaglobulinemia as determined by the Investigator.
* For Atacicept Drug Holiday Group only: Aspartate aminotransferase, alanine aminotransferase or alkaline phosphatase level >2.5 × upper limit of normal (ULN) or total bilirubin >1.5 x ULN. If the participant has a known history of Gilberts (history of isolated increase in total bilirubin without increase in liver transaminases), contact the Medical Monitor for further discussion.
* For Atacicept Drug Holiday Group only: Administration of live and live-attenuated vaccinations within 30 days prior to enrollment.
* For Atacicept Drug Holiday Group only: History or current diagnosis of any demyelinating disease such as, but not restricted to, multiple sclerosis (MS) or optic neuritis (ON)
* Active clinically significant viral, bacterial or fungal infection, or any major episode of infection requiring hospitalization or treatment with parenteral anti-infectives within 4 weeks prior to enrollment, or completion of oral anti-infectives within 2 weeks prior to enrollment, ora history of recurrent infections (ie, 3 or more of the same type of infection in a 12-month rolling period). Vaginal candidiasis, onychomycosis and genital or oral herpes simplex virus considered by the Investigator to be sufficiently controlled are not exclusionary.
* Atacicept Drug Holiday Group only: If the participant is undergoing current treatment for latent tuberculosis infection (LTBI), they must have received at least 4 continuous weeks of an appropriate LTBI treatment prior to screening without evidence of re-exposure to be eligible for this study. If on LTBI treatment at the Screening visit, the participant will be expected to complete an appropriate LTBI treatment regimen to remain in the trial

Prohibited medications:

* Use of systemic corticosteroids (including oral budesonide) or immunosuppressive medications (eg, MMF, azathioprine, cyclophosphamide, hydroxychloroquine) for the treatment of IgAN within 2 months prior to Screening
* For glucocorticosteroids (GCS), "Systemic" is defined as oral, rectal or injectable (intravenous or intramuscular) routes of administration, Other routes of administration are allowed, including intra-articular, inhaled, topical, ophthalmic, optic and intranasal
* Use of B-cell-directed biologic therapies including belimumab, rituximab, ocrelizumab within 12 months of screening
* Use of other biologics (eg, anti-TNF, abatacept, anti-IL-6) and investigational biologics for the treatment of IgAN within 6 months of screening

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events observed during the dosing period | Baseline until end of study up to week156
  Patient incidence of reported Adverse Events (AEs)

SECONDARY OUTCOMES:
To evaluate the effect of atacicept on change in proteinuria | Baseline until end of study up to week156
  Changes in proteinuria based on UPCR (Urine Protein Creatinine Ratio) and UACR (Urine Albumin-Creatinine Ratio) on spot urine.
To evaluate the effect of atacicept on the change in estimated glomerular filtration rate (eGFR) using serum creatinine and cystatin C, respectively | Baseline until end of study up to week156
  Changes in estimated glomerular filtration rate (eGFR) based on serum creatinine and cystatain C, respectively
To evaluate the effect of atacicept on hematuria | Baseline until end of study up to week156
  Hematuria level based on blood on urine dipstick
To evaluate the effect of atacicept on serum galactose-deficient IgA1 (Gd-IgA1) levels | Baseline until end of study up to week156
  Changes in serum Gd-IgA1 levels

CONTACTS AND LOCATIONS:
Overall Officials: Zeeshan Khawaja, Study Director — Vice President, Clinical Development
Locations (1):
- Vera Therapeutics, Brisbane, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vera Therapeutics, Inc Company Website — http://www.veratx.com